CLINICAL TRIAL: NCT03692936
Title: Computed Tomography Derived Fractional Flow Reserve for Coronary Hemodynamic Ischemia Noninvasive Assessment (CT-FFR-CHINA)
Brief Title: Computed Tomography Derived Fractional Flow Reserve for Coronary Hemodynamic Ischemia Noninvasive Assessment
Acronym: CT-FFR-CHINA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Beijing heart century medical technology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Bin Lu, Professor and Director of the Department of Radiologic Imaging, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: CNCCD
Record Dates: First submitted 2018-09-30; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Computed Tomography Derived Fractional Flow Reserve (CT-FFR) is a noninvasive method for evaluating the hemodynamic significance of coronary artery lesions by using coronary CT Angiography (CCTA) as opposed to invasive FFR examination under invasive coronary angiography. The purpose of the CT-FFR-CHINA study is to verify that the diagnostic performance of hemodynamically significant lesions by CT-FFR is superior than routine anatomic evaluation of diameter stenosis using CCTA alone using invasive FFR as the reference standard, exclusively in Chinese population.

DETAILED DESCRIPTION:
Numerous studies have demonstrated high diagnostic accuracy of CCTA to detect and exclude coronary artery disease (CAD). One main limitation of CCTA, however, is a tendency to overestimate the severity of coronary artery stenosis against invasive coronary angiography (ICA). On the other hand, FFR, invasively measured under ICA, is recognized as the current gold standard in determination of coronary artery lesions due to improved long-term clinical outcomes when revascularization is guided by FFR instead of ICA. Moreover, prior studies indicated unreliable relationships between detection of obstructive anatomic coronary artery stenoses defined by CCTA and hemodynamically significant lesions by invasive fractional flow reserve (FFR).

Recent advances in artificial intelligence and computational modeling techniques now permit construction of a 3-dimensional model of coronary arteries visible from CCTA images and computation of FFR anywhere in the entire 3D model noninvasively. Several prior prospective, multicenter studies have reported promising results for the diagnostic performance of CT-FFR using invasive FFR as the reference standard. However, the diagnostic performance of CT-FFR in Chinese population is not clear. Therefore, we hereby designed the CT-FFR-CHINA study to determine the hemodynamically significant lesions, exclusively in Chinese subjects. It is a prospective and multi-center trial with a total of 326 subjects enrolled at 4 Chinese centers.

ELIGIBILITY:
Inclusion Criteria:

* General Criteria:

  * Stable and unstable angina pectoris or secondary evaluation of stenosis after acute MI
  * Age > 18 years
  * Able to provide signed informed consent

CCTA inclusion criteria:

* At least one stenosis with diameter stenosis of 30%-90% by visual estimate
* Reference vessel size > 2 mm in stenotic segment by visual estimate

Exclusion Criteria:

* General Criteria:

  * Ineligible for diagnostic intervention or FFR examination
  * Myocardial infarction within 72 hours
  * Severe heart failure (NYHA≥III)
  * S-creatinine>150µmol/L or GFR<45 ml/kg/1.73m2
  * Allergy to contrast agent or adenosine
  * Factors that might substantially impact the CCTA image quality, e.g, frequent atrial premature beat or atrial fibrillation

Angiographic exclusion criteria:

* The interrogated stenosis is caused by myocardial bridge
* Ostial lesions less than 3 mm to the aorta
* Poor angiographic image quality precluding contour detection
* Severe overlap of stenotic segments
* Severe tortuosity of target vessel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with coronary artery disease admitted for coronary angiography due to high risk of significant coronary stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity of CT-FFR compared with CCTA | 7days
  In comparison to CCTA, sensitivity and specificity of CT-FFR determine whether a subject has hemodynamically-significant coronary artery lesions using binary outcomes when compared to invasive FFR as the reference standard.

SECONDARY OUTCOMES:
accuracy, positive predictive value, negative predictive value of CT-FFR compared with CCTA | 7days
  In comparison to CCTA, accuracy, positive predictive value, negative predictive value of CT-FFR to determine whether a subject has hemodynamically-significant coronary artery lesions using binary outcomes when compared to invasive FFR as the reference standard
the area under the receiver operating characteristic curve of CT-FFR compared with CCTA | 7days
  In comparison to CCTA, the area under the receiver operating characteristic curve of CT-FFR in determining whether a subject has hemodynamically-significant coronary artery lesions using binary outcomes when compared to invasive FFR as the reference standard

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Chao-Yang Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital, Beijing, Beijing Municipality
  - Qi Lu Hospital, Shan Dong University, Jinan, Shandong
  - Sir Run Run Shaw Hospital, Zhe Jiang University School of Medicine, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Gao Y, Zhao N, Song L, Hu H, Jiang T, Chen W, Zhang F, Dou K, Mu C, Yang W, Fu G, Xu L, Li D, Fan L, An Y, Wang Y, Li W, Xu B, Lu B. Diagnostic Performance of CT FFR With a New Parameter Optimized Computational Fluid Dynamics Algorithm From the CT-FFR-CHINA Trial: Characteristic Analysis of Gray Zone Lesions and Misdiagnosed Lesions. Front Cardiovasc Med. 2022 Mar 22;9:819460. doi: 10.3389/fcvm.2022.819460. eCollection 2022. PMID 35391840
- [Derived] Gao Y, Zhao N, Song L, Hu F, Mu C, Gao L, Cui J, Yin D, Yang W, Xu B, Lu B. Diastolic versus systolic coronary computed tomography angiography derived fractional flow reserve for the identification of lesion-specific ischemia. Eur J Radiol. 2022 Feb;147:110098. doi: 10.1016/j.ejrad.2021.110098. Epub 2021 Dec 14. PMID 34974364